CLINICAL TRIAL: NCT04551534
Title: A First-In-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Oral Doses of DNL201 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL201 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-B-0001
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — 2-methyl-2-(3-methyl-4-((4-(methylamino)-5-(trifluoromethyl)pyrimidin-2-yl)amino)-1H-pyrazol-1-yl)propanenitrile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DNL201 (Experimental): Part 1: Single-ascending dose cohorts; Part 2: Multiple-ascending dose cohorts (10 days); Part 3: Additional multiple-dose cohort (10 days)
  Interventions: Drug: DNL201
- Placebo (Placebo Comparator): Part 1: Single-ascending dose cohorts; Part 2: Multiple-ascending dose cohorts (10 days); Part 3: Additional multiple-dose cohort (10 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL201 — Oral dose(s)
  Arms: DNL201
Drug: Placebo — Oral dose(s)
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single- and multiple-ascending oral dose study conducted in three parts.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index 18.5 to 35.0 kg/m², inclusive, and body weight of at least 50.0 kg at screening
* In good health, determined by no clinically significant findings from medical history, physical examination, and vital sign measurements
* Women of non-childbearing potential and men using contraceptive measures

Key Exclusion Criteria:

* History of clinically significant hematological, renal, pancreatic, gastrointestinal, hepatic, cardiovascular, metabolic, endocrine, immunological, allergic disease, or other major disorders
* History of asthma, chronic obstructive pulmonary disease, or emphysema
* Clinically significant neurologic disorder
* History of stomach or intestinal surgery or resection
* History of malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs), and discontinuations due to TEAEs | Up to 20 days
PK parameter: Maximum observed concentration (Cmax) of DNL201 in plasma | Up to 10 days
PK parameter: Time to maximum observed concentration (Tmax) of DNL201 in plasma | Up to 10 days
PK parameter: The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of DNL201 in plasma (single dosing only) | Up to 10 days
PK parameter: Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) of DNL201 in plasma | Up to 10 days
PK parameter: The area under the concentration-time curve over a dosing interval (AUC0-τ) of DNL201 in plasma (multiple dosing only) | Up to 10 days
PK parameter: Apparent terminal elimination half-life (t1/2) of DNL201 in plasma | Up to 10 days

SECONDARY OUTCOMES:
Concentration of DNL201 in cerebrospinal fluid (CSF) (following selected single and multiple doses) | Up to 10 days
The pharmacodynamics of DNL201 in whole blood as measured by the percent change from baseline in pS935 | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Study Director — Denali Therapeutics Inc.
Locations (1):
- Clinical Site(s), Dallas, Texas, United States

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102